CLINICAL TRIAL: NCT01718639
Title: Randomized, Controlled, Single-blind, Three-way Crossover Clinical Investigation to Evaluate Safety and Efficacy of IQP-LH-101 in Postprandial Heartburn
Brief Title: Safety and Efficacy of IQP-LH-101 in Postprandial Heartburn
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: InQpharm Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: INQ/012512
Record Dates: First submitted 2012-10-25; First posted 2012-10-31 (Estimated); Last update posted 2013-03-11 (Estimated); Status verified 2013-03

CONDITIONS: Postprandial Heartburn

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- IQP-LH-101 tablet (Active Comparator): 4 chewable tablets to be chewed thoroughly before swallowing
  Interventions: Device: IQP-LH-101 tablet
- IQP-LH-101 liquid (Active Comparator): 2 liquid sachets to be emptied into the mouth and consumed.
  Interventions: Device: IQP-LH-101 liquid
- Placebo (Placebo Comparator): 1 tablet to be swallowed with water.
  Interventions: Other: Placebo

INTERVENTIONS:
Device: IQP-LH-101 tablet — Oral medical device in the form of a chewable tablet
  Arms: IQP-LH-101 tablet
Device: IQP-LH-101 liquid — Oral medical device in the form of a liquid
  Arms: IQP-LH-101 liquid
Other: Placebo
  Arms: Placebo

SUMMARY:
This study is a randomized, placebo-controlled, single-blind, three-way crossover clinical trial to evaluate safety and efficacy of IQP-LH-101 (tablet form and liquid form) in postprandial heartburn.

The null hypothesis is that there is no difference between IQP-LH-101 and the placebo in terms of efficacy for postprandial heartburn treatment.

ELIGIBILITY:
Inclusion Criteria:

* Post-prandial heartburn (e.g. after a high-fat meal) in at least 2 months prior to the study (at least 2 times a week)
* Not receiving prescribed treatment for heartburn, reflux or upper gastrointestinal disorders
* Written informed consent is a prerequisite for subject enrollment.

Exclusion Criteria:

* Gastrointestinal bleeding within 12 months prior to the study
* Difficulty swallowing (dysphagia)
* History of or symptoms suggestive of Zollinger-Ellison syndrome, oesophageal or gastric malignancy, gastric or duodenal ulcer, pernicious anaemia, Barrett's oesophagus or systemic sclerosis
* Participation in other studies within the last 30 days prior to entry or during the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2012-10; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Difference in time to both onset of soothing and onset of cooling after intake of investigational product between study arms | Measured up to 30 minutes
  The subject will be provided with a stopwatch started by the study staff at the time of investigational product application

SECONDARY OUTCOMES:
Duration of time until the first perception of recurring heartburn symptoms after intake of investigational product | Up to 4 hours
  The subject will be instructed to stop the stopwatch provided at first perception of recurring heartburn symptoms.
Evaluation of efficacy | Up to 4 hours per crossover
  The subjects evaluate the efficacy of the device under investigation (global scaled eval-uation with "very good", "good", "moderate" and "poor").
Adverse events | Up to 4 weeks
  The investigator will assess and document in the CRF any adverse events, device effects and device deficiencies.

CONTACTS AND LOCATIONS:
Locations (1):
- Weißenseerweg 111, Berlin, State of Berlin, Germany